CLINICAL TRIAL: NCT05097729
Title: Transcranial Magnetic Stimulation to Enhance Cortical Hippocampal Functional Connectivity as a Novel Means for Relieving Chronic OA Pain
Brief Title: rTMS for Relieving Chronic OA Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary data in chronic back pain patients showed no benefits of the treatment; we did not further pursue the same treatment in osteoarthritis patients.
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Apkar Apkarian, Director Center for Translational Pain Research, Director Center of Excellence for Chronic Pain and Drug Abuse Research, Professor of Neuroscience, Anesthesia, PM&R, Northwestern University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00214446
Record Dates: First submitted 2021-10-18; First posted 2021-10-28 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Chronic Pain; Osteo Arthritis Knee
MeSH Terms: conditions — Chronic Pain | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will receive all the 3 modalities of stimulation in a randomized order. Each round is composed by 5 daily sessions of stimulation. Participants will have a second MRI only after Modality one (hippocampal).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Stimulation Modality 1 (Experimental): Repetitive TMS will be applied at 100% resting motor threshold intensity to a region of interest located in the parietal cortex, that will be determined based on its connectivity with the hippocampus.
  Interventions: Device: Transcranial Magnetic Stimulation
- Stimulation Modality 2 (Sham Comparator): Parameters will be identical to the modality 1, except that the coil will be flipped over.
  Interventions: Device: Transcranial Magnetic Stimulation
- Stimulation Modality 3 (Active Comparator): The stimulation will be delivered over the motor cortex contralateral to the predominant painful region, i.e., right motor cortex stimulation if left knee pain. The stimulation intensity will be set at 80% of the resting motor threshold.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The brain stimulation can be delivery using different devices; in this project a MagPro X100 stimulator connected to a MagPro Cool-B65 liquid-cooled butterfly coil (MagVenture A/S, Farum, Denmark) will be used. Resting motor threshold (M1-rTMS) will be determined during the visit 1 or visit 2 and used along all visits. The rTMS pulse sequences and intensities used are all within the published safety guidelines
  Other Names: TMS

SUMMARY:
In this study the investigators aim to examine the effects of Transcranial Magnetic Stimulation (TMS) on hippocampal network connectivity and pain levels in individuals with pain due to knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) pain is one of the most prevalent causes of chronic pain worldwide. Symptoms can last from months to a lifetime, severely impacting patients' quality of life. New strategies - including non-invasive brain stimulation techniques - have shown promise for sustained pain relief, yet evidence on their reliability and efficacy is limited. Apkarian et. al have previously shown that the dorsal hippocampus plays a central role in pain analgesia; thus, the study aim is to test whether non-invasively enhancing dorsal hippocampus activity is a useful new strategy for pain relief in knee OA patients. This study will recruit 35 patients with chronic OA pain for > 6 months. Each participant will receive 3 rounds of different treatment modalities in a cross-over manner. Each treatment modality will consist of 5 daily consecutive rTMS sessions followed by a 2-weeks wash-out period. Questionnaires will be completed prior to and following each intervention, and after each treatment round. Participants will be trained to use a pain electronic application (smartphone-based tool to rate pain intensity and mood on NRS scales, as well as indicate rescue medication use, developed in our lab). They will be asked to use this application for 7-10 days prior to the first round of intervention and during the study duration.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 6 months of knee pain on a daily basis;
* male or female with no racial or ethnic restrictions;
* 18 to 75 years old;
* average knee pain intensity > 4/10 at study entry;
* must be able to read, understand, and sign consent form;
* generally healthy.
* able to use the PainApp

Exclusion Criteria:

* rheumatoid arthritis, ankylosing spondylitis, acute vertebral fractures,
* Chronic neurologic conditions, e.g., Parkinson's
* other severe medical diseases;
* pregnancy;
* positive urinary screen for any recreational drugs,
* opioids use;
* use of anticoagulants (low dose ASA allowed);
* history of gastric ulcer; renal insufficiency or congestive heart failure,
* contraindication to MRI,
* contraindication to TMS; including history of seizure/epilepsy*
* Any medical condition that in the investigator's judgment may prevent the individual from completing the study or put the individual at undue risk;
* In the judgment of the investigator, unable or unwilling to follow protocol and instructions.
* Diagnosis of major depression.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Pain ratings (Numeric Rating Scale) | Pain ratings immediately after each rTMS modality and effects after the end of stimulation round (1 week).
  The primary efficacy outcomes are the effects of the rTMS modalities on pain app ratings.

SECONDARY OUTCOMES:
Pain trajectories | 1 to 12 weeks (end of the study)
  Individual pain trajectories will be analyzed to assess rTMS effects with greater temporal granularity.
Brain biomarkers and psychological indicators of rTMS effects and pain relief | 1 to 12 weeks (end of the study)
  Test for objective mechanistic brain correlates (using functional magnetic resonance imaging - fMRI) for treatment efficacy. Specific regions of interest (ROI) involved in the hippocampal network will be studied.
Adverse events | 1 to 12 weeks (end of the study)
  Incidence of adverse events will be reported for after each rTMS session.The frequency and severity of adverse effects will be compared between each rTMS modality.
Global impression of change | 1 to 12 weeks - after each rTMS round.
  Global impression of change (PGIC): this questionnaire reflects a patient's belief about the efficacy of treatment. Although widely used in chronic pain clinical trials, PGIC's validity has not been formally assessed. PGIC is a 7 point scale depicting a patient's rating of overall improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes